CLINICAL TRIAL: NCT06649071
Title: Clinical Classification and Imaging Markers in Patients of Obesity
Status: Enrolling by invitation | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yan Bi, Clinical Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: OB2024
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Obesity; fMRI; Clinical Classification
MeSH Terms: conditions — Obesity | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — DNA and mRNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Naturalistic observation — Naturalistic observation

SUMMARY:
This is an observational study to explore the etiology and clinical classification in patients with obesity and to achieve personalized treatment.

DETAILED DESCRIPTION:
In this project, individuals with obesity and control individuals were recruited and followed up every year. Clinical neuropsychological scores, olfactory function tests, and functional magnetic resonance imaging (fmri) were performed to describe the brain function characteristics under different odor stimulation in fasting and after eating, and to explore the pathogenesis and clinical classification of obese patients. The correlation analysis between imaging analysis values and clinical laboratory data, neuropsychological scores and olfactory behavior scores was performed to explore indicators related to cognitive decline and provide new insights into the etiology and classification of obese patients. Combined with clinical evaluation and imaging examination, the changes of cognitive behavior and brain structure and function in obese patients were followed up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI≥28kg/m2
* Aged 18-65 years of both sexes, right-handed
* At least 6 years of education
* Patients agreed and signed the informed consent

Exclusion Criteria:

* Fewer than 6 years of education
* Left-handedness
* Dementia
* Acute metabolic complications such as diabetic ketoacidosis
* Hyperglycaemic hyperosmolar state and hypoglycaemic coma within the previous 3 months; history or presence of neurological or psychiatric disorders;
* Presence of hypothyroidism;
* History of malignancy, or severe kidney or liver dysfunction.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a dynamic prospective cohort study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Brain imaging features in patients with obesity by fMRI | From 2024 to 2028
  total brain volume, grey matter volume, white matter volume,cerebrospinal fluid volume, and nuclear bulk volume by MRI-derived normalized measures. All patients underwent odor-induced task fMRI on a 3.0T MR scanner with 222 volumes for task fMRI and 230 volumes for resting-state fMRI.
Biomarkers of patients with obesity by blood sample | From 2024 to 2028
  Diagnostic biomarkers, predictive biomarkers, and prognostic biomarker in patients with obesity by blood sample
Clinical classification of patients with obesity | From 2024 to 2028
  Based on the exploration of the unique brain imaging and biomarkers in patients with obesity, the clinical classification of obese patients was carried out.
Prevention and intervention strategies for obesity based on clinical classification | From 2024 to 2028
  According to the clinical classification of obesity investigated in our previous study, personalized prevention and treatment strategies are designed to effectively slow down or reverse the obesity disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, M.D., Ph.D., Study Director — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Department of Endocrinology, Endocrine and Metabolic Disease Medical Center, Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No